CLINICAL TRIAL: NCT05138913
Title: Prospective Randomized Controlled Study on Arthroscopic Treatment Combine With TXA for Elbow Stiffness
Brief Title: Arthroscopic Treatment Combine With TXA for Elbow Stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YLu
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Tranexamic Acid; Elbow Stiffness
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Arthroscopic treatment with TXA injection
  Interventions: Drug: TXA
- Control group (Placebo Comparator): Arthroscopic treatment with normal saline injection
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: TXA — After the arthroscopic operation was completed, a local TXA injection was performed
  Arms: Study group
Drug: Saline — After the arthroscopic operation was completed, a local saline injection was performed
  Arms: Control group

SUMMARY:
This study is a prospective randomized controlled study of different arthroscopic treatments for elbow stiffness combined with tranexamic acid(TXA) injection. The patients with stiffness were randomly divided into groups before the operation. After the arthroscopic operation was completed, they were divided into a local TXA injection group and a control group (normal saline) to perform additional operations for reduction of hemorrhage. In different time periods, the quantitative and qualitative indicators including pain, functional score, range of motion, level of Hemoglobin, the circumference of the limb 10cm above and below the elbow, amount of hemorrhage, etc. were compared between groups at the same time period to evaluate the difference in the effect of arthroscopic treatment combined with TXA on the treatment of reduction of hemorrhage. Determine the effectiveness of TXA.

ELIGIBILITY:
Inclusion Criteria:

Clinically diagnosed patients with elbow stiffness Young and middle-aged patients aged 18 to 60 with failed nonoperated treatment Voluntarily accept randomized controlled grouping, cooperate with treatment and follow up patients No other comorbidities or medical diseases affect the surgical patients -

Exclusion Criteria:

Elderly people older than 60 years old and patients younger than 18 years old With severe comorbidities or medical diseases affect the surgical patients

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score | baseline-6 months postoperatively
  A score used to evaluated the elbow function

SECONDARY OUTCOMES:
Visual analogue scale | baseline-6 months postoperatively
  A score used to evaluated the pain
Circumference of upper extremity | baseline-6 months postoperatively
change of hemoglobin | baseline-6 months postoperatively
range of motion | baseline-6 months postoperatively
  flexion, extension, pronation and supination of elbow

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No